CLINICAL TRIAL: NCT07040995
Title: FASTTRACK - Facilitated Access to Optimized Treatment and Clinical Follow-Up for Elderly Patients by the Internal Medicine Heart Failure Outpatient Clinic - a Randomized Multicenter Prospective Study
Brief Title: Facilitated Access to Optimized Treatment and Clinical Follow-Up for Elderly Patients by the Internal Medicine Heart Failure Outpatient Clinic - a Randomized Multicenter Prospective Study
Acronym: FASTTRACC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to unforseen changes in the flow of patients with heart failure, the study interfered with another ongoing study and was therefore withdrawn
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2024-04155-01
Record Dates: First submitted 2024-09-05; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
Keywords: older adults; elderly; heart failure; follow-up; internal medicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Patients in the control arm will receive follow-up post-discharge at the internal medicine heart failure outpatient clinic within 2 weeks. They will thereafter be referred to their primary care physician
- Interventional arm (Active Comparator): Patients in the interventional arm will receive follow-up post-discharge at the internal medicine heart failure outpatient clinic within 2 weeks. They will thereafter receive further follow-up at the internal medicine heart failure outpatient clinic on-demand for the following 6 months
  Interventions: Other: Swift follow-up

INTERVENTIONS:
Other: Swift follow-up — Swift and structured follow-up on-demand for 6 months at a disease-specific outpatient clinic following hospitalization for heart failure among older adults
  Arms: Interventional arm

SUMMARY:
Research problem and specific questions:

Due to lack of resources and an increasingly heavy burden placed on the primary care system, most of heart failure (HF) patients don´t receive a swift follow-up according to guideline recommendations. Our study aims to investigate if a structured and swift follow-up at a dedicated internal medicine HF out-patient clinic (IM-HF)) for older adults with HF post hospital discharge, can improve the quality of life and reduce mortality and re-hospitalization compared to current standard with follow-up within the primary care.

Data and method:

The study will be performed as a prospective, randomized controlled trial (RCT) at two sites. All patients older than 70 years admitted to a ward with new onset or chronic HF will be invited to participate. After discharge, all patients will be invited to a re-visit to the IM-HF within 2 weeks, and will thereafter be randomized to either continued follow-up on-demand at the IM-HF or within the primary care. Outcomes will be self-reported quality of life, number of days alive and out of hospital, time to death or re-hospitalization and adherence to guideline-directed medical therapy. Data collection will be performed by means of nurse-led interviews, blood sampling and review of medical records. By employing a RCT-design with a well-defined population, intervention, control and outcome, this study aims to provide high-quality evidence that could influence clinical practice.

Societal relevance and utilization:

The study is expected to give valuable insight into the effects of early and structured follow-up for older adults with HF and could improve the standard of care and lead to improved quality of life and reduced risks of re-hospitalization and mortality. Through multidisciplinary teams and cooperation with patients associations the study aspires to be evidence based and patient centered. The start-up and implementation of the study is expected during the following years and may have important implications for the care of older adults with HF.

Plan for project realization:

The study aims to start at the IM-HF at two sites in 2025 with a research nurse with a 50% position at each site. About 12 patients fulfilling the inclusion criteria are discharged from the hospital wards each week and we expect an inclusion rate of 4 patients/week. The study is expected to go on for 3.5 years.

DETAILED DESCRIPTION:
FASTTRACC - Facilitated AccesS To Optimized TReAtment and CliniCal follow-up for elderly patients by the internal medicine heart failure outpatient clinic - a randomized multicenter prospective study

1. Abbreviations

   HF - heart failure, GDMT - guideline directed medical therapy, DAOH - days alive and out-of-hospital, CRT - cardiac resynchronisation therapy, ICD - implantable cardiac defibrillator, IM-HF - internal medicine heart failure outpatient clinic, DIM - department of internal medicine, POCUS - point-of-care ultrasound
2. Background

   Heart failure (HF) among older patients (more than 70 years of age) is one of the most common causes for hospital admission and re-admission.1 It is not only associated with increased mortality exceeding most malignant diseases, but also with a great amount of suffering and low quality of life for the patient, with repeated hospitalizations and inability to perform activities of daily life. HF also exerts a substantial financial burden on the healthcare system mostly driven by the high-rate of re-hospitalizations that accounts for more than 70% of the total HF health care cost.2,3 Thirty-day readmission rates are reported to be as high as 22-25% 4,5 and mortality risk increases for each subsequent readmission.3 Most of these patients are elderly and burdened by several co-morbidities rendering them ineligible for advanced HF treatment such as device therapy (CRT/ICD) or mechanical support. Following hospital discharge, a majority of HF patients are referred to their primary care provider for clinical follow-up and treatment optimization.6 Due to lack of resources and an increasingly heavy burden placed on the primary care system, most of these patients don't receive their follow-up until 1-2 months after hospitalization for an acute episode of HF, at which time many have already been re-admitted to the hospital.7 This practice is not in line with current guidelines that recommend early and frequent follow-up after HF hospitalization following the STRONG-HF trial. STRONG-HF studied an intensive treatment strategy of rapid up-titration of guideline-directed medication therapy (GDMT) and close follow-up after an HF admission and showed reduced symptoms, improved quality of life, and reduced the risk of 180-day all-cause death or HF readmission compared with usual care.8,9 However, as impressive and powerful the effects of the STRONG-HF trial were; the mean age of study participants were 63 years and less than 1700 patients were included from 14 countries and 87 hospitals during more than four years. This can, of course, partly be explained by the COVID-19 pandemic but still raises the question of STRONG-HF's applicability in the everyday real-world clinical setting with an elderly HF-population with multiple co-morbidities who are unlikely to tolerate the aggressive strategy enlisted in STRONG-HF. This creates an evidentiary vacuum for the elderly HF-patients and their response to intensified GDMT that our study intends to fill.

   Almost half of all HF re-admissions are estimated to be a result of suboptimal transitional care i.e., the vulnerable phase between discharge from the hospital and initiation and continuity of care in the outpatient setting.10,11

   In a Cochrane report from 2017, nurse home visits and disease management clinics (DMC) were the only interventions in transitional care services that showed a reduction in mortality, as well as a reduced rates of re-admission for HF. Furthermore, these services were also shown to reduce health care system costs.12 Adherence to guidelines is therefore affected. The Evolution-HF study by Savarese et al found that less than 25% of discharged HF patients reach the target dose for several established heart failure drugs.13 Even in a specialized setting, the adherence to guidelines has been reported to be even lower.14

   Independently, but in consistency with the Evolution-HF study, a dedicated outpatient clinic focused on an early and structured follow-up of patients recently hospitalized for HF was initiated at the Department of Internal Medicine (DIM) Malmö at Skåne University Hospital in early 2024, with the tentative name of internal medicine heart failure outpatient clinic (IM-HF). A similar clinic is already present since 2018 at the affiliated hospital in Lund. The purpose of the IM-HF is to offer all patients hospitalized for an acute episode of HF, regardless of co-morbidities and advanced age, a quick follow-up within 2 weeks of discharge. At this visit, patients will meet with a team of dedicated physicians and nurses to implement and optimize guideline directed medical therapy (GDMT), monitor pertinent laboratory values (e.g., renal function, iron status), evaluation of congestion status, and provide information and education in self-care and lifestyle interventions with the ultimate objective being an increase in HF patients health-related quality of life, as well as a reduction in re-admission rates and mortality risk.
3. Overall aim This study aims to investigate the efficacy of a structured and prompt follow-up at a dedicated disease management clinic for older patients recently hospitalized for HF. Specifically, we will compare this approach to the current standard of care, which involves unspecified follow-up by the primary care providers.
4. Methods

   4.1 Work plan

   4.1.1 Project organization This study will be developed and coordinated from DIM in Malmö. The research team will be led by the main applicants (MO and JM), senior consultants in internal medicine and cardiology, respectively, at Region Skåne/Lund University. 40% of their research time (currently 50% research time of full time). The research group consists of 4 postdoctoral fellows, 1 PhD students and 2 study nurses. A collaboration with the patient organisation Riksförbundet Hjärt-Lung (RHL) will ensure the project's applicability and dissemination of results to a broad demographic outside of the scientific community. A representative from RHL will be invited to management group meetings when aspects of the trial importance, and patient perspective, including aspects with ethical implications, are discussed. FASTTRACC will comply with the EU regulation 536/2014 on clinical trials.

   4.1.2 Study design This study is designed as a multicenter prospective randomised study. Two sites; the IM-HF in Malmö and in Lund, will participate in the study.

   4.2 Study population: Patients ≥70 years hospitalized at the departments of internal medicine or cardiology in Malmö and Lund due to worsening symptoms of HF (both new-onset and chronic).

   Inclusion criteria:
   * Written informed consent (paper-based or digital/remote)
   * Age ≥70 years
   * Clinical diagnosis of HF
   * Follow-up after hospitalisation would otherwise be in the primary care setting

   Exclusion criteria:
   * Eligibility to advanced HF treatment such as device therapy or mechanical support
   * Intended follow-up at the Department of Cardiology (electrical cardioversion excluded)
   * Inability to give informed consent

   4.3 Intervention: Patients will be invited to a visit within 2 weeks after hospitalization. During this visit, they will undergo a comprehensive evaluation by a team of dedicated physicians and nurses. This includes implementing and optimizing GDMT, monitoring laboratory values, assessing congestion status, and providing education on self-care and lifestyle interventions. After a visit at IM-HF, patients will be randomized to either further follow-up on demand based on patients' clinical needs and need for further optimization of GDMT at the IM-HF during the following 6 months (interventional group) or standard of care in the primary care setting with a written referral to the primary care provider with recommendations of a structured medical optimization with scheduled visits at their discretion (control group). Both groups will be followed by phone interview by a study nurse as well as a written referral with blood samples at 1-, 3- and 6-months. Randomization will be performed in balanced blocks of fixed size. Patients will be randomized in the designated randomization module in the REDCap Electronic Data Capture system.

   4.4 Endpoints

   Primary endpoints:
   * "Percent Days alive and out of hospital" (%DAOH), defined as the percent of days the patient is alive and not hospitalized during the study period
   * Change in Quality of Life assessed by Kansas City Cardiomyopathy questionnaire (KCCQ) from baseline

   Secondary endpoints:
   * Time to the combined endpoint of 1-year mortality and 30-day re-admission for HF
   * Adherence to GDMT (assessed via phone interview by study nurse)

   Exploratory endpoints:
   * Time to 1-year mortality (assessed via registries)
   * Time to 30-day readmission (assessed via registries)

   4.5.1 Data collection

   Vital parameters and anthropometric measurements will be collected on site at inclusion and at the first re-visit. At follow-up at 1-, 3- and 6-months, vital parameters will be registered by means of self-monitoring. All patients will be offered the possibility of self-monitoring by using "Digital Hands" (Siemens Healthineers). Cognitive function will be assessed by Montreal Cognitive Assessment at study enrolment. Point-of-care-ultrasound (POCUS) will be carried out where appropriate. Blood samples collected will be stored in a biobank. An application to Kvalitetsregister, vårddatabaser och beredning (KVB) will be submitted and thereafter background medical history including echocardiography or POCUS will be obtained through chart review of electronic medical records (Melior, Siemens). Mortality will be assessed through the Causes of Death Registry and rehospitalisation will be assessed through the National Patient Registry. DAOH will be calculated based on mortality and rehospitalization data. KCCQ, GDMT and blood samples will be assessed at 1-,3- and 6-month follow-up. Blood samples will be analysed for iron status, changes in renal function and in NT-proBNP-levels, and at a later stage also for proteomics and metabolomics.

   4.5.2 Chart review at baseline:

   Patients fulfilling the inclusion/exclusion criteria will be subjected to manual chart review, which will be done consecutively. Baseline will be the date of discharge from hospital. The chart review will be performed according to prespecified definitions, and the following data will be collected:

   • Age at baseline

   • Sex
   * Length in centimeters (may be retrieved from earlier hospitalizations)
   * Weight in kilograms at discharge (as close to baseline as possible, ±3 weeks is acceptable)
   * Body mass index (derived from length and weight)
   * Comorbidities (Admission and Discharge notes will be scrutinized, any mentioning or ICD-10 code will be noted, results as yes/no)
   * Functional impairment - none / home care / nursing home

     - Activities of daily living before hospitalization
   * Clinical frailty scale (derived from chart review)
   * Chronic cognitive impairment
   * Echocardiography
   * If no echocardiography available, has cardiac POCUS been performed (yes/no)? If yes:

     - What was the estimated ejection fraction? Mildly, moderately or severely reduced?

     - Heart failure with preserved ejection fraction (HFpEF)?

     - Right ventricular failure?
   * NT-proBNP, iron status and renal function at discharge
   * Ceiling of care decision

     * None / no ICU escalation / no cardio-pulmonary resuscitation

   4.5 Laboratory analysis

   Blood samples will be drawn at inclusion, at the re-visit to the IM-HF and at 1-, 3- and 6-month follow-up and will then be stored in a biobank. When further funding has been secured, analysis of proteomics and metabolomics is planned.

   4.6 Statistical analysis

   Cox proportional hazards regression models will be used to estimate hazard ratios and 95% confidence intervals (CIs) for the intervention effect on time to mortality or re-hospitalization, adjusting for potential confounders. The proportional hazards assumption will be assessed using graphical methods and statistical tests. Subgroup analyses will be conducted to explore potential effect modification by relevant covariates, such as age, sex, baseline ejection fraction, or comorbidities. Interaction tests will be performed to assess the significance of intervention-covariate interactions.

   4.6.1 Estimated sample size and power

   The adjusted sample size per group was calculated to 257 participants per arm (total n=514), based on an assumed effect size of 0.2, an alpha level of 0.05, and a power of 80%. This calculation accounts for a non-responder rate of 10% and a drop-out rate of 20%.

   4.7 Time plan

   Assuming a weekly inclusion rate of n=4 (2 participants per site and week) the study duration is estimated to be 2.5 years, with an additional one year of follow-up.

   Preparation phase (0-3 months) - Month 1-2: Application to the ethics review board. Registration of the trial at ClinicalTrials.gov. Development and testing of data collection tools (RedCap).

   - Month 2-3: Training of study staff in the study protocol and data collection procedures. Establishment of logistics.

   Inclusion/intervention phase (4-30 months)
   * Month 4-30: Patient recruitment at an average rate of 2 patients/week/hospital (4 patients in total/week).
   * Month 4-36: Follow-up for patients according to study protocol. Planned return visits at 1-14 days, 8-21 days, and follow-up at 1, 3 and 6 months.

   Data collection and analysis phase (4-48 months)
   * Month 4-48: Continued data and sample collection. Data entry and validation in RedCap.
   * Month 37-48: Statistical analysis. Results and reporting phase (48-54 months)
   * Month 48-54: Compilation of results. Publication of results in scientific journals and presentation at conferences. Summary report to patient organizations and participants.

   5.0 Ethical considerations

   Approval from the Swedish Ethical Review Authority was received on the 14th of August 2024. The study will comply with the Helsinki Declaration of Ethical Research. Informed consent will be obtained from all participants, providing comprehensive information about the study´s purpose, procedures, risks, and benefits, and affirming participants right to withdraw without repercussions. A thorough risk-benefit assessment will be conducted to evaluate potential harms and benefits. Maintaining equipoise will be emphasized, ensuring unbiased treatment allocation and avoiding coercion toward a particular study arm. Data integrity and confidentiality will be upheld through secure storage (RedCap) and adherence to ethical guidelines for data management.

   6.0 Feasibility

   The existing healthcare infrastructure´s capacity to accommodate the study requirements is deemed satisfactory. Also, the ability to recruit and enroll eligible participants within the specified timeframe is considered to be satisfactory given that approximately 14 patients per week are discharged from the internal medicine wards in Malmö and Lund. This suggests that even a modest attendance rate of 28% would meet the requirements for recruitment adequately. However, we anticipate a higher attendance rate due to the potential self-perceived benefits for the patients involved. Loss to follow-up is considered insignificant for the hard endpoints of mortality and hospitalization, given the extensive accuracy and coverage provided by the Swedish registers pertaining to these outcomes. Patient adherence to the assigned follow-up protocol will be monitored at visits and via phone interviews by study nurses. For other outcomes, such as self-reported health-related quality of life and adherence to GDMT, we presume that conducting phone interviews offers a viable alternative to in-clinic visits for this particularly fragile cohort, thereby mitigating inconvenience.

   7.0 Clinical perspectives

   Rehospitalizations and low self-reported quality of life are common among patients with heart failure. In this study, we focus on the group of older adults (≥70 years) that have been discharged after hospitalization for heart failure, and that otherwise would have been referred to their primary care physician for follow up. In this vulnerable group, we aim to investigate whether follow-up visits in close proximity to a HF hospitalization at a designated medical clinic can improve the health-related quality of life, as well as reduce rehospitalization and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (paper-based or digital/remote)
* 70 years or older
* Clinical diagnosis of HF
* Follow-up after hospitalization would otherwise be in the primary care setting

Exclusion Criteria:

* Eligibility to advanced HF treatment such as device therapy or mechanical support
* Intended follow-up at the Department of Cardiology (electrical cardioversion excluded)
* Inability to give informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | From enrollment and at 1-, 3- and 6-months
  Quality of Life assessed by Kansas City Cardiomyopathy questionnaire, KCCQ
Days Alive and Out-of-hospital | From enrollment and 1 year forward
  Percentage of Days Alive and Out-of-hospital (%DAOH)

SECONDARY OUTCOMES:
1-year mortality and 30-day re-admission | From enrollment and 1 year forward for mortality. From enrollment and 30 days forward for re-admission
  Time to the combined endpoint of 1-year mortality and 30-day re-admission for heart failure
Adherence to guidline-directed medical therapy (GDMT) | From enrollment and at 1-, 3- and 6-months
  Adherence to guidline-directed medical therapy (GDMT)

OTHER OUTCOMES:
Time to 30-day re-admission | 30 days
  Time to 30-day re-admission
Time to 1-year mortality | 1 year
  1-year mortality

CONTACTS AND LOCATIONS:
Overall Officials: Amra Jujic, PhD, Study Director — Institution of Clinical Sciences, Lund University, Malmö; Hannes Holm-Isholth, MD, PhD, Study Director — Institution of Clinical Sciences, Lund University, Malmö

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Greene SJ, Butler J, Albert NM, DeVore AD, Sharma PP, Duffy CI, Hill CL, McCague K, Mi X, Patterson JH, Spertus JA, Thomas L, Williams FB, Hernandez AF, Fonarow GC. Medical Therapy for Heart Failure With Reduced Ejection Fraction: The CHAMP-HF Registry. J Am Coll Cardiol. 2018 Jul 24;72(4):351-366. doi: 10.1016/j.jacc.2018.04.070. PMID 30025570
- [Background] Mebazaa A, Davison B, Chioncel O, Cohen-Solal A, Diaz R, Filippatos G, Metra M, Ponikowski P, Sliwa K, Voors AA, Edwards C, Novosadova M, Takagi K, Damasceno A, Saidu H, Gayat E, Pang PS, Celutkiene J, Cotter G. Safety, tolerability and efficacy of up-titration of guideline-directed medical therapies for acute heart failure (STRONG-HF): a multinational, open-label, randomised, trial. Lancet. 2022 Dec 3;400(10367):1938-1952. doi: 10.1016/S0140-6736(22)02076-1. Epub 2022 Nov 7. PMID 36356631
- [Background] Savarese G, Kishi T, Vardeny O, Adamsson Eryd S, Bodegard J, Lund LH, Thuresson M, Bozkurt B. Heart Failure Drug Treatment-Inertia, Titration, and Discontinuation: A Multinational Observational Study (EVOLUTION HF). JACC Heart Fail. 2023 Jan;11(1):1-14. doi: 10.1016/j.jchf.2022.08.009. Epub 2022 Sep 7. PMID 36202739
- [Background] Van Spall HGC, Rahman T, Mytton O, Ramasundarahettige C, Ibrahim Q, Kabali C, Coppens M, Brian Haynes R, Connolly S. Comparative effectiveness of transitional care services in patients discharged from the hospital with heart failure: a systematic review and network meta-analysis. Eur J Heart Fail. 2017 Nov;19(11):1427-1443. doi: 10.1002/ejhf.765. Epub 2017 Feb 24. PMID 28233442
- [Background] Phelan D, Smyth L, Ryder M, Murphy N, O'Loughlin C, Conlon C, Ledwidge M, McDonald K. Can we reduce preventable heart failure readmissions in patients enrolled in a Disease Management Programme? Ir J Med Sci. 2009 Jun;178(2):167-71. doi: 10.1007/s11845-009-0332-6. Epub 2009 May 1. PMID 19408042
- [Background] Hernandez AF, Greiner MA, Fonarow GC, Hammill BG, Heidenreich PA, Yancy CW, Peterson ED, Curtis LH. Relationship between early physician follow-up and 30-day readmission among Medicare beneficiaries hospitalized for heart failure. JAMA. 2010 May 5;303(17):1716-22. doi: 10.1001/jama.2010.533. PMID 20442387
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Skibelund AK; ESC Scientific Document Group. 2023 Focused Update of the 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2023 Oct 1;44(37):3627-3639. doi: 10.1093/eurheartj/ehad195. No abstract available. PMID 37622666
- [Background] Laveau F, Hammoudi N, Berthelot E, Belmin J, Assayag P, Cohen A, Damy T, Duboc D, Dubourg O, Hagege A, Hanon O, Isnard R, Jondeau G, Labouree F, Logeart D, Mansencal N, Meune C, Pautas E, Wolmark Y, Komajda M. Patient journey in decompensated heart failure: An analysis in departments of cardiology and geriatrics in the Greater Paris University Hospitals. Arch Cardiovasc Dis. 2017 Jan;110(1):42-50. doi: 10.1016/j.acvd.2016.05.009. Epub 2016 Dec 21. PMID 28017276
- [Background] Liljeroos M, Stromberg A. Introducing nurse-led heart failure clinics in Swedish primary care settings. Eur J Heart Fail. 2019 Jan;21(1):103-109. doi: 10.1002/ejhf.1329. Epub 2018 Oct 19. PMID 30338881
- [Background] Dharmarajan K, Hsieh AF, Lin Z, Bueno H, Ross JS, Horwitz LI, Barreto-Filho JA, Kim N, Bernheim SM, Suter LG, Drye EE, Krumholz HM. Diagnoses and timing of 30-day readmissions after hospitalization for heart failure, acute myocardial infarction, or pneumonia. JAMA. 2013 Jan 23;309(4):355-63. doi: 10.1001/jama.2012.216476. PMID 23340637
- [Background] Bueno H, Ross JS, Wang Y, Chen J, Vidan MT, Normand SL, Curtis JP, Drye EE, Lichtman JH, Keenan PS, Kosiborod M, Krumholz HM. Trends in length of stay and short-term outcomes among Medicare patients hospitalized for heart failure, 1993-2006. JAMA. 2010 Jun 2;303(21):2141-7. doi: 10.1001/jama.2010.748. PMID 20516414
- [Background] Norton C, Georgiopoulou VV, Kalogeropoulos AP, Butler J. Epidemiology and cost of advanced heart failure. Prog Cardiovasc Dis. 2011 Sep-Oct;54(2):78-85. doi: 10.1016/j.pcad.2011.04.002. PMID 21875507
- [Background] Stewart S, Jenkins A, Buchan S, McGuire A, Capewell S, McMurray JJ. The current cost of heart failure to the National Health Service in the UK. Eur J Heart Fail. 2002 Jun;4(3):361-71. doi: 10.1016/s1388-9842(01)00198-2. PMID 12034163
- [Background] Greene SJ, Fonarow GC, Vaduganathan M, Khan SS, Butler J, Gheorghiade M. The vulnerable phase after hospitalization for heart failure. Nat Rev Cardiol. 2015 Apr;12(4):220-9. doi: 10.1038/nrcardio.2015.14. Epub 2015 Feb 10. PMID 25666406